CLINICAL TRIAL: NCT03029624
Title: Subcutaneous Tibial Nerve Stimulation for Urgency Urinary Incontinence
Brief Title: eCoin Tibial Nerve Stimulation for OAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valencia Technologies Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111-3175
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Results first posted 2020-11-27 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-11

CONDITIONS: Urgency Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Treatment Arm (Experimental): Treatment Arm receives implanted eCoin device and therapy is turned ON.
  Interventions: Device: eCoin

INTERVENTIONS:
Device: eCoin — Patients are implanted with active implantable device called eCoin. eCoin is turned ON in order to deliver neuromodulation therapy.

SUMMARY:
The study is a single arm, prospective study of the safety and effectiveness of the Valencia Technologies eCoin System to stimulate the tibial nerve for the treatment of patients with refractory urgency urinary incontinence.

DETAILED DESCRIPTION:
This trial is a single arm, prospective study of the safety and effectiveness of eCoin tibial nerve stimulation in 25 subjects with refractory overactive bladder as defined by the American Urological Association.. The eCoin neuromodulation device will be implanted subcutaneously in the right or left leg of patients with urgency urinary incontinence. After a 4 week implant healing period, subjects will have their devices activated (turned ON). After 3 months of device therapy (occurring 4 months post-implant), the primary endpoint will be assessed. It is anticipated that subjects will reach the full therapeutic effect at approximately 3 months of therapy. Subjects will be followed for an additional 9 months to assess the safety of maintenance stimulation therapy with fewer sessions occurring during this time interval.

ELIGIBILITY:
Inclusion Criteria:

1. Women and men 18 years and older.
2. Diagnosis of overactive bladder with urgency urinary incontinence or mixed urge and stress incontinence with a predominant urgency component, for at least 6 months (self-reported).
3. Individual has at least four urgency incontinence episodes on a three-day voiding diary with at least one episode per 24 hour time period
4. Individual with urinary frequency, defined as an average of greater than or equal to 8 times/24 hours (ie. a total of greater than or equal to 24 micturitions on a 3 day diary)
5. Individual is unresponsive to, inadequately responsive to, or intolerant of behavioral, rehabilitation, and pharmacologic therapy.
6. Individual is able to give his or her written, informed consent.
7. Individual is mentally competent and able to understand all study requirements.
8. Individual is willing and able to complete a 3-day voiding diary and quality of life questionnaire.
9. Individual is without pharmacological treatment of overactive bladder (antimuscarinics and beta-3 agonists) for 2 weeks prior to screening.
10. The individual demonstrates a positive nerve integrity test.

Exclusion Criteria:

1. Individual has predominantly stress urinary incontinence
2. Individual has clinically significant bladder outlet obstruction.
3. Individual has clinically significant pelvic organ prolapse.
4. Individual has abnormal post void residual (i.e., greater than 150 cc).
5. Individual has clinically significant urethral stricture disease or bladder neck contracture
6. Individual has an active urinary tract infection at time of enrollment.
7. Individual has recurrent urinary tract infections defined as 4 or more UTI's per year.
8. Individual has morbid obesity.
9. Individual has had positive urine cytology or diagnosis of bladder or prostate cancer.
10. Individual has neurogenic bladder dysfunction.
11. Individual is taking an alpha-blocker for benign prostatic hyperplasia.
12. Individual is pregnant or intends to become pregnant during the study.
13. Patient is breast feeding or is less than 9-month post-partum.
14. Individual has the presence of urinary fistula, bladder stone, or interstitial cystitis.
15. Individual has uncontrolled diabetes mellitus.
16. Individual has a cardiac pacemaker or implanted defibrillator.
17. Individual has been previously treated with sacral nerve stimulation.
18. Individual has been treated with onabotulinumtoxinA in the previous 9 months prior to enrollment.
19. Individual has been treated with percutaneous tibial nerve stimulation within the previous 12 weeks prior to enrollment.
20. Individual requires regular Magnetic Resonance Imaging for other health care conditions. (ASK)
21. Individual has a clotting or bleeding disorder; antiplatelet and anticoagulant therapy may be continued or held at the discretion of the investigator
22. Individual has a clinically significant peripheral neuropathy.
23. Individual is neutropenic or immunocompromised.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2018-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon English, MD, Principal Investigator — Urology Associates; Scott MacDiarmid, MD, Principal Investigator — Alliance Urology Specialists
Locations (7):
- United States (4):
  - The Clark Center for Urogynecology, Newport Beach, California
  - UnityPoint Clinic, Waterloo, Iowa
  - Alliance Urology Specialists, Greensboro, North Carolina
  - The Institute for Female Pelvic Medicine & Reconstructive Surgery (FPM Institute), Allentown, Pennsylvania
- New Zealand (3):
  - Urology Associates, Christchurch
  - Roundhay Medical Centre, Nelson
  - Tauranga Urology Research Ltd, Tauranga

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaaki B, English S, Gilling P, Meffan P, Lucente V, MacDiarmid S, Clark M, Sen SK. Six-Month Outcomes of Reimplantation of a Coin-Sized Tibial Nerve Stimulator for the Treatment of Overactive Bladder Syndrome With Urgency Urinary Incontinence. Female Pelvic Med Reconstr Surg. 2022 May 1;28(5):287-292. doi: 10.1097/SPV.0000000000001105. Epub 2022 Sep 22. PMID 35536667

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and enrolled from April 2017 to September 2017 (i.e. 5 months). The study took place at 7 urology/urogynecology clinics across the United States and New Zealand.
Pre-assignment Details: Participants were required to complete a 2-week washout of all overactive bladder medications prior to baseline. After passing screening and baseline criteria, patients were enrolled. As this is a single-arm study, once participants were enrolled they were assigned to the intervention (eCoin).
Groups:
- eCoin: Treatment arm receives implanted eCoin device and therapy is turned ON.
  eCoin: Patients are implanted with active implantable device called eCoin. eCoin is turned ON in order to deliver neuromodulation therapy.
Period: Overall Study
Arm/Group | eCoin
Started (Recruited) | 46
Primary Endpoint (3 Months) | 44
Completed | 41
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 1
Not completed — MRI need | 2

BASELINE CHARACTERISTICS:
Population: Baseline analyses includes the baseline information for enrolled and implanted participants. Data on 3 participants were imputed per protocol.
Arm/Group | eCoin
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.39 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 45
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  New Zealand | 20
  United States | 26
Urinary incontinence [Mean (Standard Deviation); unit: episodes/day] | 5.9 (3.1)
Urgency urinary incontinence [Mean (Standard Deviation); unit: episodes/day] | 5.2 (2.9)
No. OAB medication at screening [Count of Participants; unit: Participants] | 9
No. OAB medication history [Count of Participants; unit: Participants] | 46
Incontinence Quality of Life (I QoL) score [Mean (Standard Deviation); unit: score on a scale] — Total score reported. Range from 0-100. Lower score indicates poor quality of life, higher score indicates better quality of life.
  score on a scale | 45.39 (20.4)

OUTCOME MEASURES:

1. Primary Outcome: Incontinent Episodes
Description: The change in number of incontinence episodes from baseline to three months post-activation.
Time Frame: Baseline to three months post-activation.
Population: Intent-to-treat
Measure: Median (Standard Deviation); unit: episodes/day
Arm/Group | eCoin
Number analyzed (Participants) | 46
episodes/day | -3.0 (2.9)

2. Secondary Outcome: System and Procedure Related AEs
Description: Number of System and Procedure Related Adverse Events from implantation to one month post-implantation.
Time Frame: Implantation to one month post-implantation.
Population: Intent-to-treat
Measure: Number; unit: Adverse Events
Arm/Group | eCoin
Number analyzed (Participants) | 46
Adverse Events | 20

3. Secondary Outcome: MAEs
Description: Number of all Major Adverse Events from baseline to 3 months post-activation.
Time Frame: Baseline to 3 months post-activation.
Population: Intent-to-treat
Measure: Number; unit: Adverse Events
Arm/Group | Treatment Arm
Number analyzed (Participants) | 46
Adverse Events | 3

4. Secondary Outcome: Percentage of Responders
Description: Percentage of Responders, defined as participants who experienced a 50% or greater reduction in UUI after 3 months of treatment
Time Frame: 3 months after activation
Measure: Count of Participants; unit: Participants
Arm/Group | eCoin
Number analyzed (Participants) | 46
Participants | 32

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from enrollment through 6 months after implantation.
Description: The safety population consisted of all eligible and enrolled participants. AEs were graded at the study centers as mild, moderate, or sever; serious or not serious; classified as related or unrelated; and classified as causing or not causing study termination. The Data Safety and Monitoring Board reviewed all AEs to confirm relatedness.
Arm/Group | eCoin
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 3/46
Other Adverse Events (participants affected / at risk) | 16/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | eCoin (N=46)
Cellulitis Secondary to Ankle Wrap (Infections and infestations) | 1 (1) — One participant experienced cellulitis secondary to an ankle wrap that was part of the specified wound care but with no involvement of the incision or implant site. Cellulitis resolved with intravenous antibiotics.
Hip Bursitis & Edema (Musculoskeletal and connective tissue disorders) | 1 (1) — Participant presented with limp and pain determined to be related to hip bursitis and edema, which were noted at screening.
Pneumonia (Infections and infestations) | 1 (1) — Participant contracted pneumonia determined to be unrelated to the device and resolved with treatment
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | eCoin (N=46)
Mild swelling, bruising, discomfort (General disorders) | 3 (4)
Possible incision site infection (Infections and infestations) | 2 (2)
Blister secondary to ankle wrap (Skin and subcutaneous tissue disorders) | 4 (4)
Moderate implant site discomfort, swelling, pain, bruising (General disorders) | 5 (5)
Stimulation pain (Product Issues) | 1 (1)
Device migration about 1 cm posterior (Product Issues) | 1 (1)

LIMITATIONS AND CAVEATS:
This was a small study with a nonrandomized design and no control group. Studies in larger populations may clarify the factors associated with responders. The initial study period was short at only 3 months, and should be investigated further for durability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-19): https://cdn.clinicaltrials.gov/large-docs/24/NCT03029624/Prot_SAP_000.pdf